CLINICAL TRIAL: NCT04918615
Title: PROMISE-BIF ：A Prospective, Multicenter, Randomized Controlled Trial to Compare the Efficacy and Safety of Sirolimus Coated Balloon Catheter With Paclitaxel Coated Balloon Catheter for the Treatment of De Novo Coronary Bifurcated Lesions
Brief Title: Compare Sirolimus Coated Balloon Catheter With Paclitaxel Coated Balloon Catheter in De Novo Coronary Bifurcated Lesions
Acronym: PROMISE-BIF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-IC-040
Record Dates: First submitted 2021-06-04; First posted 2021-06-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
Keywords: drug coated balloon catheter; coronary bifurcation lesion
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sirolimus coated balloon catheter (Experimental): Manufacturer: Shanghai MicroPort Medical Group Co, Ltd.
  Interventions: Procedure: PCI
- Paclitaxel coated balloon catheter (Active Comparator): Manufacturer: Liaoning Yinyi Biotechnology Co., Ltd
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — Patients in experimental group will undergo PCI with drug coated balloon catheter to treat the side branch of the coronary bifurcation lesion.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Microport sirolimus drug coated balloon catheter for the treatment of coronary bifurcation lesions.

DETAILED DESCRIPTION:
PROMISE-BIF is a prospective, multicenter, randomized controlled, non-inferior clinical trial, which would enroll about 234 participants. All participants will undergo PCI with sirolimus drug coated balloon catheter or paclitaxel drug coated balloon catheter and be followed-up to 24 months.

The Target Lesion defined as the true bifurcation, include the main branch and side branch lesion.

The bifurcation lesions were classified by Medina (1.1.1, 1.0.1, and 0.1.1). The image data will be analyzed and evaluated independently by a third-party imaging laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female ages 18-80 years old
* Participants with myocardial ischemia, stable or unstable angina pectoris, old myocardial infarction, or Stabled myocardial infarction (occurred more than 7 days before enrollment, including non-ST elevation and ST elevation myocardial infarction)
* Participants are are eligible to undergo any type of coronary revascularization surgery, such as balloon angioplasty, stenting, and coronary artery bypass grafting (CABG);
* Participants Can understand the trial's purpose, voluntarily participate and acknowledge all the risks and benefits, providing written informed consent and are willing to accept invasive radiographic during the follow-up period.
* Angiography confirmed as De novo bifurcation lesion, the stenosis rate of side branch (diameter) ≥70％
* Suitable for PCI and the side branch lesions is not expected to stent implantation, and no DCB treatment for the main branch. If a stent is implanted into the main-branch, it's usually necessary to perform a final balloon kissing on the two branches
* Up to 2 vessels that need to be treated, total intended treat lesions' amount will not exceed 3
* At most one primary bifurcation lesion that needs treatment (including Medina classification 1.1.1, 1.0.1, 0.1.1), ostium stenosis degree (diameter) ≥70% (visual);
* Patients are suitable for PCI and side branch is not expected to implant a stent, the main branch will not apply drug coated balloon; the main branch will implant a stent, usually the main branch and side branch will have Kissing Balloon Inflation
* The side branch is pre-dilated successfully, no C or upper grade dissection, no tear or other complications occurred, residual stenosis ≤50%, TIMI3
* The reference diameter of the target lesion side branch is 2.0~4.0 mm, the length of the lesion in side branch is ≤38 mm, and the length of the lesion in main branch is ≤70 mm

Exclusion Criteria:

* Any AMI occurred within 1 week before operation
* Unstable arrhythmias, such as high-risk ventricular premature beats, ventricular tachycardia
* severe heart failure (above NYHA IV) or Left ventricular ejection fraction (LVEF) <30% (ultrasound or left ventricular angiography)
* Renal function insufficiency: Serum creatinine >177μmol/L; Or undergoing hemodialysis;
* definite hemorrhagic tendency, antiplatelet and anticoagulant therapy contraindication and unable to anticoagulant therapy;
* PCI planned within 1 year
* Have a history of peptic ulcer or gastrointestinal hemorrhage in the past 6 months; Have a history of cerebrovascular accidents (stroke) such as cerebral hemorrhage, cerebral infarction in the past 6 months;
* allergic to contrast agent, paclitaxel, and rapamycin and its derivatives
* Has been diagnosed as advanced cancer and other serious diseases, lifespan are expected less than 12 months or hard to complete the 12-month follow up;
* Patients who are considered to have poor compliance and cannot complete the trial in accordance with requirements; Or other reasons that considered by the investigator, it be unsuitable to enroll the participant;
* Be participating in any other clinical trials, or have participated in clinical trials of other drugs or medical devices before being selected but have not reached the timeline of the primary endpoint;
* Female who are pregnant or breastfeeding (women who may become pregnant must undergo a pregnancy test within 7 days before the baseline surgery)；Or have fertility plan/can not have adequate contraception during the study period
* Three vessel disease and all the vessels need revasculization
* Left main and its bifurcation lesions;
* thrombus in the bifurcation lesion, or tortuose lesion that the balloon catheter will not pass through;
* Side branch lesion segment of target lesion is a total occlusion lesion
* side branch is severely calcified, and cannot be pre-dilated or dilated while do kissing balloon inflation;
* Target lesion (including main branch and branch) is in-stent re-stenosis
* Dissection above grade C or residual stenosis >50% after pre-dilation of the target lesion branch vessel disease or double kissing balloon dilation;
* Two or more non-target lesions that need to be treated, the non-target lesion cannot be processed before the target lesion or the treatment fails;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Diameter Stenosis (DS) of side branch | 9 months
  Stenosis of lumen diameter of lesion segment of the side branch

SECONDARY OUTCOMES:
Late lumen loss (LLL) of side branch | 9 months
  late lumen loss of lesion segment of the side branch

OTHER OUTCOMES:
Immediate Success Endpoint | 7 days
  Immediate Success Endpoint including Technical success, Lesion success and Procedural success.
  Technical success defined as the success of the study device in reaching the target lesion branch vascular lesions, dilatating and retracting successfully with residual stenosis of the branch vessel lesion ≤30%(visual inspection); Lesion success defined as the main and branch vessels of the target lesion residual stenosis Residual stenosis ≤ ≤30%, furthermore blood flow is TIMI 3 (visual inspection) after treatment with any interventional method Procedural success defined as the absence of device-related composite end point events during the hospitalization period (up to 7 days after surgery) on the basis of Lesion success.
DoCE | 30 days, 6 months, 9 months, 12 months, 24 months post-procedure
  Defined as a composite of cardiac death, target vessel-related MI, or ischemia-driven side branch lesion revascularization events at 30 days, 6 months, 9 months and 12 months
PoCE | 30 days, 6 months, 9 months, 12 months, 24 months post-procedure
  Defined as a composite rate of all cause death, all MI or any revasculariztion at 30 days, 6 months, 9 months, and 12 months
Death | 30 days, 6 months, 9 months, 12 months, 24 months post-procedure
  Cardiac, Vascular, Non-cardiovascular related
Myocardial infarction | 30 days, 6 months, 9 months, 12 months, 24 months post-procedure
  Target vessel related, Non-target vessel related
Target lesion Revascularization | 30 days, 6 months, 9 months, 12 months, 24 months post-procedure
  Lesion revascularization in main branch, side branch or both, ischemic driven or non-ischemic driven
Target vessel Revascularization | 30 days, 6 months, 9 months, 12 months, 24 months post-procedure
  Ischemia-driven , Not ischemia-driven
Any coronary revascularization | 30 days, 6 months, 9 months, 12 months, 24 months post-procedure
  Ischemia-driven , Not ischemia-driven
Thrombotic events | 30 days, 6 months, 9 months, 12 months, 24 months post-procedure
  ARC defined: acute, subacute, late
AE & SAEs rate | 30 days, 6 months, 9 months, 12 months, 24 months post-procedure
side branch re-stenosis rate | 9 months
  the proportion of patients with re-stenosis in the side branch, stenosis degree >50%
main branch re-stenosis rate | 9 months
  the proportion of patients with re-stenosis in the main branch, stenosis degree >50%
In-segment late loss of the main branch (mm) | 9 months
  The minimum lumen diameter (MLD) immediately after stent implantation was subtracted from the MLD at follow-up
In-segment Stenosis degree of the main branch (%) | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of the PLA Northern Theater Command, Shengyang, Liaoning, China